CLINICAL TRIAL: NCT04771520
Title: Phase 2 Study of Avapritinib in Patients With CKIT or PDGFRA Mutation-Positive Malignant Solid Tumors
Brief Title: Avapritinib for the Treatment of CKIT or PDGFRA Mutation-Positive Locally Advanced or Metastatic Malignant Solid Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0439; NCI-2021-00702 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0439 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-02-08; First posted 2021-02-25 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Clinical Stage IV Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage IVA Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage IVB Gastroesophageal Junction Adenocarcinoma AJCC v8; Locally Advanced Malignant Solid Neoplasm; Locally Advanced Melanoma; Locally Advanced Primary Malignant Central Nervous System Neoplasm; Locally Advanced Sarcoma; Metastatic Malignant Solid Neoplasm; Metastatic Melanoma; Metastatic Primary Malignant Central Nervous System Neoplasm; Metastatic Sarcoma; Pathologic Stage IV Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IVA Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IVB Gastroesophageal Junction Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IV Gastroesophageal Junction Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IVA Gastroesophageal Junction Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IVB Gastroesophageal Junction Adenocarcinoma AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8; Prognostic Stage IV Breast Cancer AJCC v8; Stage IIIC Colorectal Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8; Stage IV Colorectal Cancer AJCC v8; Stage IV Lung Cancer AJCC v8; Stage IVA Colorectal Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Colorectal Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8; Stage IVC Colorectal Cancer AJCC v8
MeSH Terms: conditions — Neoplasm Metastasis; Melanoma; Sarcoma; Colorectal Neoplasms; Lung Neoplasms | interventions — avapritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (avapritinib) (Experimental): Patients receive avapritinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Avapritinib

INTERVENTIONS:
Drug: Avapritinib — Given PO
  Other Names: (S)-1-(4-fluorophenyl)-1-(2-(4-(6-(1-methyl-1Hpyrazol-4-yl)pyrrolo[2,1-f][1,2,4]triazin-4-yl)piperazin-yl)pyrimidin-5-yl)ethan-1-amine; AYVAKIT; BLU-285; CS3007; PDGFR alpha/KIT Mutant-specific Inhibitor BLU-285

SUMMARY:
This phase II trial studies the effect of avapritinib in treating malignant solid tumors that have a genetic change (mutation) in CKIT or PDGFRA and have spread to nearby tissue or lymph nodes (locally advanced) or other places in the body (metastatic). Avapritinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Avapritinib may help to control the growth of malignant solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the objective response rate (ORR) of avapritinib in patients with pathogenic CKIT or PDGFRA activating mutation-positive malignant solid tumors, as assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or RANO criteria (as appropriate).

SECONDARY OBJECTIVES:

I. To evaluate the duration of response (DoR) to avapritinib in patients with pathogenic CKIT or PDGFRA activating mutation-positive malignant solid tumors.

II. To evaluate the disease control rate (DCR) of avapritinib in patients with pathogenic CKIT or PDGFRA activating mutation-positive malignant solid tumors.

III. To determine the safety and tolerability of avapritinib in patients with pathogenic CKIT or PDGFRA activating mutation-positive malignant solid tumors, as assessed by the National Cancer institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0.

EXPLORATORY OBJECTIVES:

I. To evaluate the overall survival (OS) of patients with pathogenic CKIT or PDGFRA activating mutation-positive malignant solid tumors receiving avapritinib.

II. To evaluate the ORR and DoR of avapritinib in patients with measurable brain or central nervous system (CNS) metastases at baseline.

III. To evaluate the progression-free survival (PFS) of patients with pathogenic CKIT or PDGFRA activating mutation-positive malignant solid tumors receiving avapritinib.

IV. To evaluate the correlation between genomic mutations and clinical outcome. V. To evaluate time on treatment (including patients treated beyond progression).

VI. To evaluate baseline genomics and circulating cell-free deoxyribonucleic acid (cfDNA) and functional analyses of variants.

OUTLINE:

Patients receive avapritinib orally (PO) once daily (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* The patient (or legally acceptable representative if applicable) provides written informed consent for the study
* >= 18 years of age on the day of informed consent signing
* Patient has a locally advanced or metastatic solid tumor and has progressed on appropriate standard therapy, has not shown clinically meaningful benefit to appropriate standard therapy, has no available standard therapy, or has declined appropriate standard therapy

  * NOTE: Specific solid tumor types include but are not limited to melanoma, breast cancer, lung cancer, gastroesophageal cancer, colorectal cancer, sarcoma, solid tumors not otherwise specified (NOS), and primary central nervous system (CNS) tumors. Patients with any other solid tumor type with the exception of gastrointestinal stromal tumor (GIST) will be eligible for enrollment in the study
* Measurable disease per the RECIST v1.1 or Response Assessment in Neuro-Oncology Criteria (RANO) criteria, as appropriate (for Cohorts 1 and 2 only). NOTE: Patients in Cohort 3 can have measurable or non-measurable disease
* Documented pathogenic CKIT activating mutation (Cohort 1) OR pathogenic PDGFRA activating mutation (Cohort 2) based on tissue-based next-generation sequencing (NGS) diagnostic test (Oncomine Comprehensive Assay [OCA] or FoundationOne CDx) OR plasma cfDNA-detected (Guardant360) pathogenic CKIT or PDGFRA activating mutation (for patients with measurable disease) or tissue or cfDNA-detected pathogenic CKIT or PDGFRA activating mutation (for patients with non-measurable disease; Cohort 3). Mutation pathogenicity will be verified by the MD Anderson Cancer Center (MDACC) Precision Oncology Decision Support (PODS) team. Acceptable CKIT/PDGFRA mutations for study eligibility are listed in Appendix E.
* Has available archival tissue for CKIT or PDGFRA mutation testing (cohort 1 and 2 only).
* White blood cell count > 2,500/uL and < 15,000/uL (within 28 days of study treatment initiation)
* Absolute neutrophil count >= 1.5 x 10^9/L (without granulocyte colony-stimulating factor support within 2 weeks of laboratory test used to determine eligibility) (within 28 days of study treatment initiation)
* Platelet count >= 75 x 10^9/L (without transfusion within 2 weeks of laboratory test used to determine eligibility) (within 28 days of study treatment initiation)
* Hemoglobin >= 9.0 g/dL (without blood transfusion within 7 days of laboratory test used to determine eligibility) (within 28 days of study treatment initiation)
* Total bilirubin =< 1.5 x upper limit of normal (ULN); if hepatic metastases are present, =< 2.0 x ULN (within 28 days of study treatment initiation)
* Aspartate transaminase (AST) and alanine transaminase (ALT) =< 2.5 x ULN; if hepatic metastases are present, =< 5.0 x ULN (within 28 days of study treatment initiation)
* Serum creatinine </= 2XULN or creatinine clearance ≥45 mL/min (within 28 days of study treatment initiation)
* Cardiac ejection fraction >/= 45% per screening echocardiogram or multigated acquisition scan
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Life expectancy >= 3 months
* Willing and able to comply with the protocol for the duration of the study including treatment and scheduled visits and examinations
* Willing to undergo biopsy as required by the study
* Females must be postmenopausal (defined as >= 45 years of age with at least 12 months of spontaneous amenorrhea) or premenopausal with documented surgical sterilization (tubal ligation, hysterectomy, bilateral salpingectomy, or bilateral oophorectomy), or evidence of non-childbearing status for women of childbearing potential (negative serum beta-human chorionic gonadotropin pregnancy test) within 3 days of study treatment initiation
* Females of childbearing potential must either abstain from heterosexual intercourse or use a highly effective method of contraception for the course of the study through 6 weeks after the last dose of avapritinib.
* Males with female partners of reproductive potential must either abstain from sexual intercourse or they and their partners must use a highly effective method of contraception when engaging in sexual intercourse for the course of the study through 30 days after the last dose of study treatment

Exclusion Criteria:

* Patients who have GIST
* Patients with tyrosine kinase inhibitor (TKI)-resistant CKIT mutation V654A or T670I
* Patient with meningeal carcinomatosis, leptomeningeal carcinomatosis, spinal cord compression, or symptomatic or unstable brain metastases. Note: Patients with stable brain metastases (defined as asymptomatic or no requirement for high-dose or increasing dose of systemic corticosteroids and without imminent need of radiation therapy) are eligible (including those with untreated brain metastases). If applicable, patients must have completed brain radiation therapy and recovered adequately from any associated toxicity and/or complications prior to eligibility assessment. For patients who have received prior radiation therapy, post-treatment magnetic resonance imaging (MRI) scan should show no increase in brain lesion size/volume
* History of documented congestive heart failure (New York Heart Association functional classification III-IV) or serious cardiac arrhythmias requiring treatment
* QT interval corrected using Fridericia's formula of > 470 msec
* Is currently participating or has participated in a study of an investigational agent or has used an investigational device within 2 weeks prior to study treatment initiation
* Prior anticancer chemotherapy, hormone therapy, immunotherapy, targeted therapy, radiation therapy, or surgery within 2 weeks prior to study treatment initiation.

  * NOTE: Patients must have recovered from all adverse events (AEs) due to previous therapies to =< grade 1 or baseline (except alopecia). Patients with Grade ≤2 neuropathy are eligible
  * NOTE: If patient received major surgery, she/he must have recovered adequately from the toxicity and/or complications from the intervention prior to study treatment initiation
* Arterial thrombotic or embolic events within 6 months prior to study treatment initiation, or venous thrombotic events within 2 weeks prior to study treatment initiation
* CTCAE >= grade 3 hemorrhage or bleeding event within 4 weeks prior to study treatment initiation
* Known risk of intracranial bleeding, or a history of intracranial bleeding
* History of cerebrovascular accident or transient ischemic attacks
* Symptomatic non-healing wound, ulcer, gastrointestinal perforation, or bone fracture
* Unstable seizures or patients that have required increase doses of anti-seizure meds in the last 4 weeks.
* History of psychotic or depressive disorder. Patients whose disorder is well controlled on a stable antipsychotic or antidepressant medication for at least 12 months prior to study entry will be eligible
* Concomitant use of a known strong cytochrome P450 (CYP)3A4 inhibitor or strong CYP3A4 inducer. The required washout period prior to study treatment initiation is 2 weeks or 5x half-life (T1/2), whichever is shortest
* Females who are pregnant or breastfeeding
* Unable to swallow and retain oral medications
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of the study treatment (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
* Known additional malignancy that is progressing or requires active treatment. NOTE: Patients with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or cervical cancer in situ that have undergone potentially curative therapy are not excluded
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | or date of death from any cause, whichever came first, assessed up to 50 months
  ORR defined as confirmed complete response (CR) or partial response (PR) from the time of study treatment initiation until disease progression as centrally assessed using the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or Response Assessment in Neuro-Oncology Criteria (RANO) criteria, as appropriate. Confirmed CR or PR will be defined as a repeat assessment performed 4 weeks (+/-3 days) after the criteria for response is first met. Will estimate ORR along with 90% confidence interval according to Clopper-Pearson method for each cohort and for specific tumor type.

SECONDARY OUTCOMES:
Duration of response (DoR) | Up to study completion (estimated 4 years)
  Determined for patients with best overall response of confirmed CR or PR (centrally assessed); DoR is defined as the number of months from the start of CR or PR (whichever response is recorded first) and subsequently confirmed to the first date of documented PD or death. Descriptive statistics will be used.
Disease control rate (DCR) | >= 16 weeks following study treatment initiation
  DCR defined as BOR of confirmed CR or PR (either of any duration) or stable disease SD >= 16 weeks following study treatment initiation. Descriptive statistics will be used.
Incidence of adverse events | Up to study completion (estimated 4 years)
  Will be measured by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Descriptive statistics will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Rodon Ahnert, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M.D. Anderson Cancer Center — http://www.mdanderson.org